CLINICAL TRIAL: NCT02536326
Title: LEPU Renal Denervation System for Resistant Hypertension in Chinese Populations
Brief Title: LEPU Renal Denervation System for Resistant Hypertension
Acronym: LEPU-RDN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-ZX-028
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- renal denervation (Experimental)
  Interventions: Device: LEPU Renal Denervation System

INTERVENTIONS:
Device: LEPU Renal Denervation System — LEPU Renal denervation system was similar to Symplicity Catheter System (Medtronic Inc.)

SUMMARY:
The purpose was to evaluate 6-month outcomes of renal denervation(RDN) for the treatment of resistant hypertension in Chinese patients in a prospective cohort study.

DETAILED DESCRIPTION:
Currently, considerable data on RDN have been obtained from Western populations, while the clinical outcomes of RDN in East Asian populations are seldom reported. Therefore, the purpose was to evaluate 6-month outcomes of RDN for the treatment of resistant hypertension in Chinese patients.In a prospective single-center cohort study, 50 Chinese patients with resistant hypertension would be recruited to undergo RDN by LEPU Renal denervation system, which was similar to Symplicity the Symplicity renal-denervation system (Medtronic). The primary effectiveness endpoint was change in systolic and diastolic blood pressure at six months as measured by office-based blood pressure assessment and 24-hour ambulatory blood pressure monitoring following therapeutic renal denervation compared to baseline. The primary safety endpoint was the incidence of Major Adverse Event (MAE) through 6 months , including severe renal artery dissection/stenosis(>60%) that required stenting or surgery, cerebrovascular accident, myocardial infarction, death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Stable medication regimen including ≥3 antihypertensive medications of different classes, including a diuretic (with no changes for a minimum of 4 weeks prior to RDN)
* 1) Office SBP and/or DBP ≥160/100 mm Hg ( ≥ 150/95 mmHg for type II diabetic patients) , 2) ABPM 24 hour mean SBP and/or DBP ≥140 and/or 90 mmHg
* Main renal arteries with ≥4 mm diameter or with ≥20 mm treatable length (by visual estimation)
* eGFR ≥45 mL/min/1.73 m2
* Written informed consent

Exclusion Criteria:

1. Clinical Exclusion Criteria:

   * Known secondary hypertension
   * Type 1 diabetes mellitus
   * Has an implantable cardioverter defibrillator (ICD) or pacemaker
   * Myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within 6 months of the screening period
   * Widespread atherosclerosis with documented intravascular thrombosis or unstable plaques
   * Has hemodynamically significant valvular heart disease
   * Pregnant, nursing, or planning to be pregnant
   * Any serious medical condition that may adversely affect the safety of the participant or the study
   * Currently enrolled in another investigational drug or device trial
2. Anatomic Exclusion Criteria

   * Renal artery stenosis (≥50%) or renal artery aneurysm in either renal artery
   * History of prior renal artery intervention including balloon angioplasty or stenting
   * Multiple renal arteries where the main renal artery is estimated to supply <75% of the kidney
   * Main renal arteries with <4 mm diameter or with <20 mm treatable length (by visual estimation)
   * Renal artery abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: Reduction of systolic blood pressure(SBP) and diastolic blood pressure(DBP) at six months as measured by office-based blood pressure assessment and ambulatory blood pressure monitoring(ABPM) compared to baseline | 6 months after RDN
2.Safety: The incidence of Major Adverse Event (MAE) through 6 months , including severe renal artery dissection/stenosis(>60%) | through 6 months

SECONDARY OUTCOMES:
Reduction in 24-h ambulatory blood pressure(ABPM) parameters | 1 month,3 months,6 months after RDN
Device or procedure related acute adverse events（Renal artery edema、mural thrombus，change in transcatheter blood pressure >20%,<20% compared to baseline、reduction of heart rate >20%） | Perioperative period
Symptomatic orthostatic hypotension, hypertensive emergency necessitating hospital admission | 1 month,3 months,6 months after RDN
Change in office SBP and DBP at 1, 3 months | 1 month, 3 months after RDN
Change in average 24-hour SBP and DBP by ambulatory blood pressure monitoring (ABPM) at 1, 3 months | 1 month, 3 months after RDN
Change in renal function at 6 months: Estimated glomerular filtration rate (eGFR) reduction >25%, 50% | 6 months after RDN

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, Doctor, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College